CLINICAL TRIAL: NCT04333459
Title: A Phase 2A, Randomized, Double-Blind Study To Evaluate The Safety And Immunogenicity Of A Hantaan Virus DNA Vaccine And A Puumala Virus DNA Vaccine, For The Prevention Of Hemorrhagic Fever With Renal Syndrome, Administered To Healthy Adult Volunteers Using The Pharmajet Stratis® Needle-Free Jet Injection Delivery Device
Brief Title: Safety and Immunogenicity of a Hantaan Virus DNA Vaccine and a Puumala Virus DNA Vaccine, For The Prevention of Hemorrhagic Fever With Renal Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: S-19-06
Record Dates: First submitted 2020-03-31; First posted 2020-04-03 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Hantaan Virus Nephropathy; Puumala Virus Nephropathy
MeSH Terms: conditions — Hemorrhagic Fever with Renal Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 - Full Dose Hataan (Active Comparator): Group 1 will be vaccinated with the "Full Dose" of HTNV DNA vaccine, 2 mg of pWRG/HTN-M(co) with 0.5 mg/each deltoid.
  Interventions: Biological: Hataan DNA Vaccine/Puumala DNA Vaccine
- Group 2 - Half Dose Hataan (Active Comparator): Group 2 will be vaccinated with the "Half Dose" of HTNV DNA vaccine, 1 mg of pWRG/HTN-M(co) with 1.0 mg/each deltoid.
  Interventions: Biological: Hataan DNA Vaccine/Puumala DNA Vaccine
- Group 3 - Full Dose Puumala (Active Comparator): Group 3 will be vaccinated with the "Full Dose" of PUUV DNA vaccine, 2 mg of pWRG/PUU-M(s2) with 1.0 mg/each deltoid.
  Interventions: Biological: Hataan DNA Vaccine/Puumala DNA Vaccine
- Group 4 - Half Dose Puumala (Active Comparator): Group 4 will be vaccinated with the "Half Dose" of PUUV DNA vaccine, 1 mg of pWRG/PUU-M(s2) with 1.0 mg/each deltoid.
  Interventions: Biological: Hataan DNA Vaccine/Puumala DNA Vaccine

INTERVENTIONS:
Biological: Hataan DNA Vaccine/Puumala DNA Vaccine — Vaccine compared in High and Lose Doses.

SUMMARY:
A randomized 4 cohort study that is comparing the data collected during the earlier phase study and to determine if immunogenicity can be retained with a 1 mg dose of Hantaan DNA vaccine.

DETAILED DESCRIPTION:
The study will enroll 4 randomized groups of 33 subjects each for a total of 132 subjects. Every subject will receive a total of 4 vaccinations. Subjects and study personnel will be blinded to the group that they are randomized to (double-blind). The study is intended to substantiate the Phase 1 results with the 2 mg dose and to also determine if immunogenicity can be retained with a 1 mg dose (for HTNV DNA vaccine).

For the 2 mg dose, each vaccination consists of 2 administrations of 1 mg (left and right deltoid) for a total of 2 mg/vaccination. For the 1 mg dose, each vaccination consists of 2 administrations of 0.5 mg (left and right deltoid) for a total of 1 mg/vaccination.

Group 1 will be vaccinated with the HTNV DNA vaccine, pWRG/HTN-M(co) at the 2 mg/vaccination dose. Group 2 will be vaccinated with the HTNV DNA vaccine, pWRG/HTN-M(co) at the 1 mg/vaccination dose. Group 3 will be vaccinated with the PUUV DNA vaccine, pWRG/PUU-M(s2) at the 2 mg/vaccination dose. Group 4 will be vaccinated with the PUUV DNA vaccine, pWRG/PUU-M(s2) at the 1 mg/vaccination dose. Each group will be vaccinated on Days 1, 29, 57 and 169. All doses will be administered with the PharmaJet Stratis device, which is FDA cleared for IM administration of vaccines. All subjects will be followed until 1 month after the last vaccination with Day 197 being the final study visit. Subjects will complete post-injection memory aids for 7 days after each vaccination.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be included in the study:

1. Healthy adult male or nonpregnant, nonlactating female, ages 18-49 (inclusive) at the time of screening
2. Have provided written informed consent before screening
3. Completion of Study Comprehension Quiz (minimum passing score of 80% with 2 attempts permitted).
4. A subject must have a valid state or government-issued photo ID (eg, driver's license, military ID, or U.S. passport) & be able to pass a background check in order to gain access to the base & participate.
5. Free of clinically significant health problems, as determined by pertinent medical history and clinical examination with ECG and laboratory assessments prior to entry into the study
6. Available and able to participate for all study visits and procedures
7. Females subjects must have had a hysterectomy or bilateral oopherectomy or must be using an effective method of contraception** from 30 days prior to the first study vaccination until 90 days after the last study vaccination.

   ** For this study, we define an effective contraceptive method as one that results in a failure rate of less than 1% per year when it is used consistently and correctly. This includes, but is not limited to, abstinence from sexual intercourse with a male partner, monogamous relationship with a vasectomized partner, bilateral tubal ligation, or intrauterine devices.
8. Female subjects who have not had a hysterectomy or bilateral oopherectomy must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours prior to each study vaccination.
9. Sexually active male participants whose partner is a woman who has not had a hysterectomy or bilateral oopherectomy and has not had a vasectomy** must agree not to father a child until 90 days after the last vaccination.

   ** performed > 1 year prior to screening
10. Women agree to not donate eggs (ova, oocytes) and male subject agrees not to donate sperm from the start of screening onwards until at least 90 days after the last vaccination.
11. Agree not to participate in another clinical trial during the study period.
12. Agree not to donate blood to a blood bank for 3 months after receiving the last study vaccine.
13. Have acceptable screening laboratories* within 90 days prior to enrollment. Refer to Appendix A for range of acceptable laboratory values. Screening laboratory values that are outside acceptable range but are thought to be due to an acute condition or due to laboratory error may be repeated once. [see Manual of Procedures (MOP)]
14. Negative HIV testing (HIV Ab / antigen 4th generation screen with reflex confirmatory RNA testing).
15. Negative hepatitis B surface antigen (HBsAg) and hepatitis C antibody testing.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. History of previous hantavirus vaccine.
2. History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions
3. Ongoing participation in another clinical trial (those continuing through Day 197 will not join other new studies until their final visit)
4. Receipt of licensed vaccines within 7 days before or after immunization (30 days for live vaccines)
5. Any use of investigational drugs or vaccines within 30 days before starting the study.
6. Ability to observe possible local reactions at the eligible injection sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art
7. Acute or chronic, clinically significant hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the investigator based on medical history, physical exam, and/or laboratory screening test
8. Pregnant or lactating female, or female who intends to become pregnant during the study period
9. Administration of immunoglobulins and/or any blood products within the 120 days preceding study entry or planned administration during the study period
10. Blood donation for human use (eg, American Red Cross or other similar blood drives) within the 56 days preceding study entry or planned administration during the study period
11. Any confirmed evidence of hepatitis B or C infection
12. Have an acute illness*, as determined by the site PI or appropriate sub-investigator, within 72 hours prior to study vaccination.

    *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol. Subjects may re-screen after an acute illness is resolved
13. Any confirmed or suspected immunosuppressive or immunodeficient condition or use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
14. Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying drugs within 6 months of study entry

    * For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day
    * Intranasal, inhaled, and topical steroids are allowed (daily inhaled steroids for treatment of asthma are NOT allowed)
15. Any chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child and intermittent non migraine headaches
16. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
17. Have any plan to have surgery between enrollment and the end of the study.
18. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
19. Have received any antiviral within 3 days of study vaccination.
20. A diagnosis of Type I or II diabetes.
21. Suspected or known current alcohol or drug abuse. Alcohol abuse defined by an alcohol intake of greater than 3 drinks a day on average for a man, and greater than 2 drinks a day on average for a woman.
22. Unwilling to allow storage and use of blood for future hantavirus-related research
23. Any other significant finding that in the opinion of the investigator would increase the risk of the individual having an adverse outcome from participating in this study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects in Group 1 that achieve seroconversion by Day 197, which is defined as a PsVNA50 titer >= 40 or at least a four-fold increase in baseline titers | 197 (+/- 2) days
  To assess the proportion of subjects in the high dose HTNV vaccine group (Group 1) that achieve immunologic seroconversion above the minimum target threshold of 80% seroconversion, after receiving 4 doses of vaccine using the PharmaJet Stratis ® device.
The proportion of subjects in Group 3 that achieve seroconversion by Day 197, which is defined as a PsVNA50 titer >= 40 or at least a four-fold increase in baseline titers. | 197 (+/- 2) days
  To assess the proportion of subjects in the high dose PUUV vaccine group (Group 3) that achieve immunologic seroconversion above the minimum target threshold of 80% seroconversion, after receiving 4 doses of vaccine using the PharmaJet Stratis ® device

SECONDARY OUTCOMES:
The proportion of subjects in Group 2 that achieve seroconversion by Day 197, which is defined as a PsVNA50 titer >= 40 or at least a four-fold increase in baseline titers | 197 (+/- 2) days
  To assess the proportion of subjects in the low dose HTNV vaccine group (Group 2) that achieve immunologic seroconversion above the minimum target threshold of 80% seroconversion, after receiving 4 doses of vaccine using the PharmaJet Stratis ® device. This secondary objective will be evaluated only if the corresponding High Dose Group primary objective shows significance
The proportion of subjects in Group 4 that achieve seroconversion by Day 197, which is defined as a PsVNA50 titer >= 40 or at least a four-fold increase in baseline titers | 197 (+/- 2) days
  To assess the proportion of subjects in the low dose PUUVV vaccine group (Group 4) that achieve immunologic seroconversion above the minimum target threshold of 80% seroconversion, after receiving 4 doses of vaccine using the PharmaJet Stratis ® device. This secondary objective will be evaluated only if the corresponding High Dose Group primary objective shows significance.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials Center, Walter Reed Army Institute of Reserach, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided